CLINICAL TRIAL: NCT00228033
Title: Calcium for the Prevention of Postpartum Depression
Brief Title: Effectiveness of Supplemental Calcium in Preventing Postpartum Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R21MH063242 (NIH); R21MH063242 (NIH); DAHBR AD-D
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2007-12

CONDITIONS: Depression; Depression, Postpartum
Keywords: Calcium; Pregnancy; Postpartum Depression; Depression
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Calcium

INTERVENTIONS:
Drug: Elemental calcium (as carbonate)

SUMMARY:
This study will evaluate the effectiveness of taking supplemental calcium while pregnant in reducing the risk of postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression is a combination of physical, emotional, and behavioral changes that occur after childbirth. The rapid drop in estrogen and progesterone levels, as well as the social and psychological changes resulting from the birth of a child, can often trigger depression in women. Common symptoms include crying, irritability, fatigue, loss of appetite, and feelings of guilt and anxiety. Women who develop postpartum depression often feel unable to care for their baby or themselves. Postpartum depression is common; it is estimated that about 10 percent of new mothers experience some symptoms of depression following delivery. Risk factors include a personal or family history of depression and a history of suffering from premenstrual dysphoric disorder (PMDD), a severe form of premenstrual syndrome (PMS). The purpose of this study is to evaluate the effectiveness of calcium supplements taken during pregnancy in reducing the likelihood of postpartum depression in women at risk for developing this condition.

Pregnant women who are at risk for developing postpartum depression will be enrolled in this study when they are between 16 to 26 weeks pregnant. All recruited women will undergo psychological testing for screening purposes. Women who are found to be depressed or suffering from other psychiatric disorders during screening will be referred to alternative treatment and will not be enrolled in this study. All participants will then be randomly assigned to receive either a calcium supplement (2 grams) or placebo on a daily basis. Treatments will continue throughout the remainder of each woman's pregnancy and for 12 weeks after she gives birth. Outcome measurements will include standardized questionnaires and psychiatric interviews to assess depression levels. If any participant exhibits significant depressive symptoms, she will be referred for psychiatric treatment. All measurements will be assessed at Weeks 26, 32 and 38 of the pregnancy, and 6 and 12 weeks after giving birth.

ELIGIBILITY:
Inclusion Criteria:

* Less than 26 weeks pregnant
* At risk for postpartum depression due to a family or personal history of depression or history of premenstrual dysphoric disorder (PMDD)

Exclusion Criteria:

* Currently depressed
* Currently taking medications for depression, bipolar disorder, or schizophrenia
* History of medication treatment for depression within 3 months of study entry
* Any of the following illnesses: diabetes, kidney disease, parathyroid disease, or untreated thyroid disease
* Currently taking a diuretic or calcium channel blocker
* Does not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238
Dates: Start 2002-04; Primary Completion 2005-12 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Score on Edinburgh Postnatal Depression Scale; measured at Weeks 6 and 12 after childbirth
Symptoms of depression; measured throughout the study with a standard psychiatric interview

SECONDARY OUTCOMES:
Calcium effects on depression; measured througout pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Hatton, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Harrison-Hohner J, Coste S, Dorato V, Curet LB, McCarron D, Hatton D. Prenatal calcium supplementation and postpartum depression; an ancillary study to randomized trial of calcium for prevention of preeclampsia. Archives of Women's Mental Health 3(41):141-146, 2001.
- [Background] Hatton DC, Harrison-Hohner J, Coste S, Dorato V, Curet LB, McCarron DA. Symptoms of postpartum depression and breastfeeding. J Hum Lact. 2005 Nov;21(4):444-9; quiz 450-4. doi: 10.1177/0890334405280947. PMID 16280561
- [Result] Hatton DC, Harrison-Hohner J, Matarazzo J, Edwards P, Lewy A, Davis L. Missed antenatal depression among high risk women: a secondary analysis. Arch Womens Ment Health. 2007;10(3):121-3. doi: 10.1007/s00737-007-0180-1. Epub 2007 Apr 16. PMID 17431740